CLINICAL TRIAL: NCT02838563
Title: Validation of a Scale of Well-Being Assessment (SIWA) in Patients With Alzheimer's Disease or a Related Disease.
Acronym: SIWA
Status: Terminated | Type: Observational
Why Stopped: no new location to open
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0441
Record Dates: First submitted 2016-07-18; First posted 2016-07-20 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-02

CONDITIONS: Well-Being
Keywords: Dementia; Alzheimer; Well-Being
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient living in nursing home: Patient with an Alzheimer Disease or related disorder living in nursing home.
  Interventions: Other: SIWA

INTERVENTIONS:
Other: SIWA — To investigate the scale reliability over time, SIWA are assessed twice, ten minutes apart. To investigate the validity of the tool, SIWA is correlated with another quality of life questionnaire (QoL-AD), a quality of health scale including an analog portion (EQ 5D), and a behavioral disorder scale (Neuropsychiatric Inventory, NPI).

SUMMARY:
Current scales are not suited to a direct measure for the elderly with cognitive disorders and are difficult to handle for the care teams. In this context, a visual analog scale was created to answer a single question "How are you feeling now, immediately?" with the help of pictograms. This study aims to assess the validity and reliability of the Scale of Well-Being Assessment (SIWA) (in french : Echelle d'Evaluation Instantanée du Bien-Etre (EVIBE)) in people with Alzheimer's disease or a related disease.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled patients must have given themselves, or through a trusted person referred to the Article L. 1111-6 of the Code of Public Health, failing thereof, by the family, or, a person maintaining close and stable ties. For adults under guardianship, permission must be given by the legal representative of the person. The research will benefit from the backing of persons Protection Committee (PPC) prior to its implementation.
* Patient living in one of the nursing home or hospital services in the project;
* Patient with Alzheimer's or a related disease

Exclusion Criteria:

* severe, progressive or unstable pathology, which may interfere with the evaluation variables;
* deafness or blindness may compromise patient assessment

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with an Alzheimer Disease or related disorder living in nursing home
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2016-01-13 (Actual); Primary Completion 2017-04-27 (Actual); Study Completion 2017-04-27 (Actual)

PRIMARY OUTCOMES:
Correlation between SIWA and an other quality of life scale (Qol-AD) | the Qol-AD is collected once. (Day 1)
  In the Qol-Ad, the patient assesses the quality of life (bad / average / good / excellent) on five areas: relationships with friends and family, concerns about finances, physical condition, mood, and an overall assessment of life quality through 13 questions.

SECONDARY OUTCOMES:
Stability over time of SIWA | The SIWA is collected twice at ten minute intervals (Day 1)
  The SIWA is a visual analogue scale for reporting the status of the patient's well-being at a specific time. On a graduated scale from 0 to 5, the caregiver should position a cursor : position from the left corresponding to the lowest feeling of well, position from the right corresponding to the highest feeling of well-being.
Correlation between SIWA and an health scale (EQ-5D) | the EQ-5D is collected once. (Day 1)
  In the EQ 5D, the patient evaluates his state of health on 5 dimensions: mobility, human autonomy, common activities, pain / discomfort and anxiety / depression based on 3 levels "no problems", "some problems" and "severe problems". Then the patient is asked to distinguish his general state of health on an analog scale from 0 (worst imaginable health state) to 100 (best imaginable health state).
Correlation between SIWA and behavioral and psychological symptom of dementia (BPSD) (NPI) | the NPI is collected once. (Day 1)
  Each of the 12 BPSD (delusions, hallucinations, agitation, depression, anxiety, excitement, apathy, disinhibition, depression, aberrant motor behavior, sleep and appetite) is evaluated from 0 to 12, depending on its frequency and severity.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Krolak-Salmon, Pr, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Centre de Recherche Clinique " Vieillissement-Cerveau-Fragilité ", Hôpital des Charpennes, Hospices Civils de Lyon, Villeurbanne, France